CLINICAL TRIAL: NCT04163913
Title: GAPS: Digital Engagement: The Impact on Subject Compliance and Satisfaction
Brief Title: Radial Medical - GAPS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-01399
Record Dates: First submitted 2019-10-24; First posted 2019-11-15 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cirvo Device (Experimental): The CirvoTM device (Figure 1) is a lightweight, mobile, active, intermittent leg compression device placed on the calf of the leg, using hook and loop (e.g. Velcro) straps in the similar manner as commercially available intermittent leg compression devices The system utilizes an electro-mechanical drive system to intermittently compress the calf from the ankle toward the knee for a duration and compression level prescribed by the physician. The level of compression delivered by the CirvoTM therapy will be in the same range as existing devices which corresponds to the type of pressure applied by a blood pressure cuff.
  Interventions: Other: Change in User interfaces of Cirvo compression device application.; Other: Change in Satisfaction in use of Cirvo device
- ActiveCare DVT (Active Comparator): A commercially available device was previously used to assess patient satisfaction with compression therapy for DVT prophylaxis as per standard of care.
  Interventions: Other: Change in User interfaces of Cirvo compression device application.; Other: Change in Satisfaction in use of Cirvo device

INTERVENTIONS:
Other: Change in User interfaces of Cirvo compression device application. — Comparison of 2 versions of the Circo user interface
Other: Change in Satisfaction in use of Cirvo device — Comparison of how satisfied patients are with the Cirvo device to a different compression device (ActiveCare)

SUMMARY:
This study will prospectively compare compliance rates between a novel FDA cleared wearable compression therapy with and without digital engagement for DVT prophylaxis in both hospital and home environments after total knee or hip arthroplasty.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, prospective, single-center study designed to evaluate compliance to CirvoTM therapy use with and without digital engagement. Historical questionnaire data with a different compression device will be compared to the same questionnaire used for the prospective cohort of up to 200 subjects. All patients prescribed compression therapy following total joint arthroscopy will be offered participation.

Subjects will receive CirvoTM compression therapy according to the standard of care protocol at NYU during or after surgery and 18 hours per day for 14 days.

1. Baseline: Following consent, participants will provide demographic, medical history and information with respect to their elective orthopedic procedure and receive training on the CirvoTM device. Participants will be randomized to either digital engagement or no digital engagement groups.
2. Post procedure: After the procedure, CirvoTM device operation will be reviewed with the participant.
3. Discharge: Any adverse events occurring during hospitalization will be reviewed, data capture on the CirvoTM app will be confirmed.
4. 14- day visit: Participants will complete a patient satisfaction questionnaire, provide information with respect to any adverse events including specific details about DVT and readmission and return the devices.
5. 30-day phone call/visit: Participants will be contacted at 30 days to answer questions about DVT's and readmissions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over the age of 18
* Undergoing elective primary total hip/knee replacement
* Planned discharge to home
* Able to train to and operate the Cirvo device with app

Exclusion Criteria:

* History of Pulmonary Embolism
* Active cancer
* BMI >40
* Current smoker
* History of a hyper-coaguable condition
* Actual or expected prolonged bedrest for >3 days
* Calf geometry on which Cirvo device does not appropriately fit (prospective cohort only)
* Known sensitivity to any of the materials used in the Cirvo device (prospective cohort only)
* Currently participating or planning to participate in any other investigational clinical evaluation during study period that may, in the opinion of the investigator, affect compliance (prospective cohort only)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change in compliance using Cirvo compression therapy | 14 day visit (+7 days)
  A sample size of 100 subjects is powered at 90% to show a difference of 10% in compliance between the 2 digital engagement cohorts. For each subject, Compliance will be calculated for each participant during the course of therapy in terms of the number of hours of actual use/number of hours of prescribed use. The number of hours will be summarized as days of use for each group.
  The means of each group will be presented. The primary endpoint is the difference in compliance between the group assigned to digital engagement versus no digital engagement with the Cirvo app. The mean difference will be compared to zero using the paired t-test

SECONDARY OUTCOMES:
Change in patient satisfaction using Cirvo compression therapy | 14 day visit (+7 days)
  A comparison between the satisfaction of CirvoTM therapy versus the historical data from comparator device use will be performed. Results of the usability questionnaire (Patient Satisfaction Intermittent Compression Devices Questionnaire) will be qualitatively summarized.
Change in staff satisfaction using Cirvo compression therapy. | 14 day visit (+7 days)
  A comparison between the satisfaction of CirvoTM therapy versus the historical data from comparator device use will be performed. Results of the usability questionnaire will be qualitatively summarized. Staff Satisfaction Intermittent Compression Devices Questionnaire will be administered.
Change in patients satisfaction using Cirvo compression therapy | 30 day visit
  A comparison between the satisfaction of CirvoTM therapy versus the historical data from comparator device use will be performed. Results of the usability questionnaire (Patient Satisfaction Intermittent Compression Devices Questionnaire) will be qualitatively summarized.

CONTACTS AND LOCATIONS:
Overall Officials: James Slover, MD, Principal Investigator — NYU Langone Health

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). Upon reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Requests should be directed to Daniel.waren@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.